CLINICAL TRIAL: NCT03137771
Title: Maintenance Systemic Therapy Versus Local Consolidative Therapy (LCT) Plus Maintenance Systemic Therapy for Limited Metastatic Non-Small Cell Lung Cancer (NSCLC): A Randomized Phase II/III Trial
Brief Title: Maintenance Chemotherapy With or Without Local Consolidative Therapy in Treating Patients With Stage IV Non-small Cell Lung Cancer
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: NRG Oncology (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NRG-LU002; NCI-2016-00849 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); NRG-LU002 (Other: NRG Oncology); NRG-LU002 (Other: CTEP); U10CA180868 (NIH)
Record Dates: First submitted 2017-04-26; First posted 2017-05-03 (Actual); Results first posted 2025-03-11 (Actual); Last update posted 2025-11-25 (Actual); Status verified 2025-02

CONDITIONS: Recurrent Non-Small Cell Lung Carcinoma; Stage IV Non-Small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Radiotherapy, Conformal; Docetaxel; Gemcitabine; Radiotherapy, Intensity-Modulated; Pemetrexed; Radiosurgery; Erlotinib Hydrochloride; pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm 1 (systemic maintenance chemotherapy) (Active Comparator): Patients may receive docetaxel IV over 60 minutes on day 1, erlotinib hydrochloride by mouth daily, or gemcitabine IV over 30 minutes on days 1 and 8. Patients with non-squamous non-small cell lung cancer may receive pemetrexed disodium IV over 10 minutes on day 1 alone or in combination with pembrolizumab IV over 30 minutes. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Docetaxel; Drug: Gemcitabine; Drug: Pemetrexed Disodium; Drug: Erlotinib Hydrochloride; Drug: Pembrolizumab
- Arm 2 (LCT + systemic maintenance chemotherapy) (Experimental): Patients undergo local consolidative therapy (LCT) over 2-5 weeks, consisting of SBRT/hypofractionated radiation to the primary tumor and metastatic sites or surgery of metastatic sites. Hypofractionated radiation using IMRT or 3D-CRT can be given in place of SBRT. Within 2 weeks after completion of LCT (3 weeks if surgery occurred), patients receive chemotherapy as in Arm 1.
  Interventions: Radiation: 3-Dimensional Conformal Radiation Therapy (3D-CRT); Drug: Docetaxel; Drug: Gemcitabine; Radiation: Intensity-Modulated Radiation Therapy (IMRT); Drug: Pemetrexed Disodium; Radiation: Stereotactic Body Radiation Therapy (SBRT); Drug: Erlotinib Hydrochloride; Drug: Pembrolizumab

INTERVENTIONS:
Radiation: 3-Dimensional Conformal Radiation Therapy (3D-CRT) — Undergo 3DCRT
  Other Names: 3-dimensional conformal radiation therapy; 3-dimensional radiation therapy; 3D CONFORMAL RADIATION THERAPY; 3D CRT; 3D-CRT; Conformal Therapy; Radiation Conformal Therapy
  Arms: Arm 2 (LCT + systemic maintenance chemotherapy)
Drug: Docetaxel — Given IV
  Other Names: Docecad; RP56976; Taxotere; Taxotere Injection Concentrate
Drug: Gemcitabine — Given IV
  Other Names: dFdC; dFdCyd; Difluorodeoxycytidine
Radiation: Intensity-Modulated Radiation Therapy (IMRT) — Undergo IMRT
  Other Names: IMRT; Intensity Modulated RT; INTENSITY-MODULATED RADIATION THERAPY; Intensity-Modulated Radiotherapy
  Arms: Arm 2 (LCT + systemic maintenance chemotherapy)
Drug: Pemetrexed Disodium — Given IV
  Other Names: Alimta; LY231514; N-[4-[2-(2-Amino-4,7-dihydro-4-oxo-1H-pyrrolo[2,3-d]pyrimidin-5-yl)ethyl]benzoyl]-L-glutamic Acid Disodium Salt
Radiation: Stereotactic Body Radiation Therapy (SBRT) — Undergo SBRT
  Other Names: SBRT; stereotactic body radiation therapy
  Arms: Arm 2 (LCT + systemic maintenance chemotherapy)
Drug: Erlotinib Hydrochloride — Given PO
  Other Names: Tarceva
Drug: Pembrolizumab — Given IV
  Other Names: Keytruda

SUMMARY:
This randomized phase II/III trial studies how well giving maintenance chemotherapy with or without local consolidation therapy works in treating patients with stage IV non-small cell lung cancer. Drugs used in maintenance chemotherapy, such as docetaxel, pemetrexed disodium, erlotinib hydrochloride, and gemcitabine work in different ways to stop the growth of tumor cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Local consolidation therapy such as radiation/stereotactic body radiation or surgery may kill cancer cells left after initial treatment. Giving maintenance chemotherapy and local consolidation therapy together may work better than maintenance chemotherapy alone in treating patients with stage IV non-small cell lung cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

Phase II

To evaluate the impact of adding local consolidative therapy (LCT) to maintenance systemic therapy versus maintenance systemic therapy alone on progression-free survival for patients with metastatic non-small cell lung cancer (NSCLC) with no evidence of progression and limited metastatic sites after first-line systemic therapy.

Phase III

To evaluate the impact of adding LCT to maintenance systemic therapy versus maintenance systemic therapy alone on overall survival for patients with metastatic NSCLC with no evidence of progression and limited metastatic sites after first-line systemic therapy.

SECONDARY OBJECTIVES:

I. To evaluate the impact of adding LCT to maintenance systemic therapy versus maintenance systemic therapy alone on in-field local failure.

II. To evaluate the impact of adding LCT to maintenance systemic therapy versus maintenance systemic therapy alone on the time to development of new lesions.

III. To evaluate the impact of adding LCT to maintenance systemic therapy versus maintenance systemic therapy alone on toxicity.

IV. To evaluate the impact of adding LCT to maintenance systemic therapy versus maintenance systemic therapy alone on duration of maintenance systemic therapy usage.

V. To evaluate the effect of adding LCT to systemic therapy in limited stage IV NSCLC on Quality of Life (QOL).

VI. To collect biospecimens and evaluate the correlation between clinical outcomes and circulating tumor DNA (ctDNA).

Patients are randomized 2:1 between the SBRT and chemotherapy vs. chemotherapy alone arms.

After completion of study treatment, patients are followed up every 3 months for 2 years, every 6 months for 3 years, then annually thereafter.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have the psychological ability and general health that permits completion of the study requirements and required follow up
* Women of childbearing potential and men who are sexually active should be willing and able to use medically acceptable forms of contraception during the trial and for up to 180 days after completion of all treatment to prevent pregnancy or fathering a child.
* Pathologically proven diagnosis of NSCLC, with metastases (stage IV disease) present prior to registration; this includes patients newly diagnosed with metastatic disease or those initially diagnosed and treated for stage I-III NSCLC who ultimately develop limited metastases. Limited metastases is defined as 3 or fewer sites of metastatic disease
* Appropriate stage for study entry based on the following diagnostic workup:

  * History/physical examination by a radiation oncologist (and a surgeon if surgery is planned) within 30 days prior to registration
  * Imaging proof of limited metastatic disease and response to therapy/stable disease, by at least diagnostic quality CT chest through the adrenals or positron emission tomography (PET)/CT within 30 days prior to registration
* Zubrod performance status 0, 1, or 2 within 30 days prior to registration
* Adequate organ and hematologic/bone marrow function within 14 days prior to registration, defined as follows:

  * Aspartate transaminase (AST) and alanine transaminase (ALT) ≤ 2.5 × upper limit of normal (ULN) or ≤ 5 × ULN with metastatic liver disease
  * Total bilirubin ≤ 1.5 × ULN
  * Absolute neutrophil count (ANC) ≥ 500 cells/mm3
  * Platelets ≥ 50,000 cells/mm3
  * Renal:
  * Creatinine ≤ 1.5 x ULN; or
  * Creatinine Clearance (CrCl) > 45 mL/min if creatinine > 1.5 x ULN (calculated CrCl based on Cockcroft-Gault equation)
* HIV-infected patients on effective anti-retroviral therapy with undetectable viral load within 6 months are eligible for this trial.
* For patients who will undergo resection of disease (if randomized to Arm 2 and dispositioned to receive surgery), adequate pre-surgical work-up for anticipated surgery, as defined by institutional guidelines.
* Negative serum pregnancy test within one week prior to registration for females of childbearing potential
* Patients must have received first-line/induction systemic therapy comprising of immunotherapy and/or platinum-based chemotherapy (at least 4 cycles or courses but less than 6, i.e. 4-5 cycles/courses), and achieved stable disease or a partial response. Though the intention is for every course/cycle to be identical in an induction regimen, Some but not all of the 4-5 cycles may omit an immunotherapy or platinum compound if the treating physician determines it is in the patient's best interest secondary to toxicity or other institutional parameter.
* For patients treated with nivolumab, ipilimumab and 2 cycles of chemotherapy, the 4-5 cycles requirement will be met by 4-5 total doses of nivolumab.
* For patients treated with nivolumab and ipilimumab, this requirement will be met by 2 doses of ipilimumab and 4-5 doses of nivolumab.
* After induction systemic therapy, patients must have a minimum of one site of disease, primary or metastasis, present for potential consolidation with local therapy. All sites of disease present after induction systemic therapy, primary and metastases (up to 3) are able to be consolidated with local therapy;
* Prior systemic therapy as part of concurrent treatment approach for previously diagnosed stage I-III NSCLC, adjuvant or neo-adjuvant therapy for stage I-III NSCLC, as adjuvant therapy for previously resected or irradiated NSCLC, or for other previous cancers is permitted
* For de novo stage IV NSCLC patients (patients with metastatic disease at first presentation), primary disease must be treatable with local therapy in the form of SBRT or hypofractionated radiation. If the primary disease is found in the peripheral or central lung parenchyma without nodal disease, for instance, SBRT may be employed at the discretion of the treating institution. If primary disease is more advanced with involvement of the mediastinum (T4 tumor, N1-N3 disease, etc.), these volumes should be technically treatable with hypofractionated radiation; surgery should only be used for metastatic tumors that can be completely resected by lobectomy, segmentectomy, or wide wedge resection.
* If primary disease in the thoracic cavity was previously treated with local therapy in the form of surgery or radiation, any new local/regional disease recurrence should be technically treatable with SBRT or hypofractionated radiation after induction systemic therapy.
* The patient or a legally authorized representative must provide study-specific informed consent prior to registration.
* Radiotherapy for patients with brain metastases prior to registration is acceptable.
* Patients with brain metastases are eligible if these lesions have been previously treated or resolved and the patients have no clinical or radiographic evidence of progression prior to registration.
* Subjects may receive palliative radiotherapy for symptomatic metastases or primary disease prior to registration provided that there is at least one other non-irradiated lesion amenable to LCT at the time of registration.

Exclusion Criteria:

* Clinical or radiologic evidence of untreated and/or progressive brain metastases prior to registration after induction systemic therapy
* Cutaneous metastasis of NSCLC
* Metastatic disease invading the esophagus, stomach, intestines, or mesenteric lymph nodes if not a candidate for surgery for these lesions
* Prior invasive malignancy (except non-melanomatous skin cancer, low or intermediate risk prostate cancer, or in situ carcinoma of breast, oral cavity, skin, or cervix) unless disease free for a minimum of one year
* Metastases located within 3 cm of previously irradiated (< 3 Gy per fraction) structures if if not a candidate for surgery for these lesions and if:

  * Spinal cord previously irradiated to > 40 Gy
  * Brachial plexus previously irradiated to > 50 Gy
  * Small intestine, large intestine, or stomach previously irradiated to > 45 Gy
  * Brainstem previously irradiated to > 50 Gy
  * Lung previously irradiated with prior V20 Gy > 35%
* Patients receiving targeted therapy (non-cytotoxic systemic therapy) for NSCLC in the first-line setting
* Patients with NSCLC who have driver mutations for which targeted therapies (non-cytotoxic, non-immunotherapy based systemic therapy including but not limited to tyrosine-kinase inhibitors) are available. Such designations would include but not be limited to treatments targeting epidermal growth factor receptor (EGFR) mutant or anaplastic lymphoma kinase (ALK) positive NSCLC.
* If a patient has progressed in previous areas of primary disease that received definitive doses of radiation, these patients would require re-irradiation in previous high dose anatomic areas and are not eligible for this study.
* Patients with malignant pleural effusions that do not resolve after first-line systemic therapy; patients with pleural effusions that have become too small for thoracentesis at the time of registration would be permitted on study, indicating a significant response to first-line systemic therapy
* Patients with more than 3 discrete locations of extra-cranial metastatic disease after first-line systemic therapy requiring more than 3 radiation/surgery plans to cover these distinct metastatic disease entities
* Acute bacterial or fungal infection requiring intravenous antibiotics at the time of registration
* Pregnancy or women of childbearing potential and men who are sexually active and not willing/able to use medically acceptable forms of contraception during treatment and for 180 days after the completion of all treatment. This exclusion is necessary because the treatment involved in this study may be significantly teratogenic. Women who are breastfeeding (and unwilling to discontinue) are also excluded
* Participation in any investigational drug study for the treatment of cancer within 4 weeks prior to registration.
* For patients who received immunotherapy during induction, patients on chronic steroids or who have active autoimmune disease for which they received systemic treatment in the previous 2 years with corticosteroids, disease modifying agents, or immunosuppressive drugs are not eligible. Replacement therapy (thyroxine, insulin or physiological corticosteroid replacement for adrenal or pituitary insufficiency) is allowed. Patients with active interstitial lung disease or who have a history of pneumonitis for which they had received glucocorticoids are not eligible
* Use of bevacizumab or other antiangiogenic therapy in first-line or planned maintenance therapy (due to potential for increased complications from local therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 218 (Actual)
Dates: Start 2017-04-07 (Actual); Primary Completion 2023-12-20 (Actual); Study Completion 2028-12 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Puneeth Iyengar, Principal Investigator — NRG Oncology
Locations (301):
- United States (296):
  - University of Alabama at Birmingham Cancer Center, Birmingham, Alabama
  - Arizona Center for Cancer Care - Gilbert, Gilbert, Arizona
  - Arizona Center for Cancer Care-Peoria, Peoria, Arizona
  - Mayo Clinic Hospital in Arizona, Phoenix, Arizona
  - Arizona Center for Cancer Care - Scottsdale, Scottsdale, Arizona
  - Mayo Clinic in Arizona, Scottsdale, Arizona
  - University of Arizona Cancer Center-Orange Grove Campus, Tucson, Arizona
  - Banner University Medical Center - Tucson, Tucson, Arizona
  - University of Arizona Cancer Center-North Campus, Tucson, Arizona
  - University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - Alta Bates Summit Medical Center-Herrick Campus, Berkeley, California
  - City of Hope Comprehensive Cancer Center, Duarte, California
  - UC San Diego Moores Cancer Center, La Jolla, California
  - Los Angeles General Medical Center, Los Angeles, California
  - USC / Norris Comprehensive Cancer Center, Los Angeles, California
  - Memorial Medical Center, Modesto, California
  - Saint Joseph Hospital - Orange, Orange, California
  - The Permanente Medical Group-Roseville Radiation Oncology, Roseville, California
  - Sutter Medical Center Sacramento, Sacramento, California
  - University of California Davis Comprehensive Cancer Center, Sacramento, California
  - Salinas Valley Memorial, Salinas, California
  - City of Hope South Pasadena, South Pasadena, California
  - Kaiser Permanente Cancer Treatment Center, South San Francisco, California
  - Saint Helena Hospital, St. Helena, California
  - Gene Upshaw Memorial Tahoe Forest Cancer Center, Truckee, California
  - Penrose-Saint Francis Healthcare, Colorado Springs, Colorado
  - UCHealth Memorial Hospital Central, Colorado Springs, Colorado
  - Porter Adventist Hospital, Denver, Colorado
  - Poudre Valley Hospital, Fort Collins, Colorado
  - Yale University, New Haven, Connecticut
  - Helen F Graham Cancer Center, Newark, Delaware
  - Beebe Health Campus, Rehoboth Beach, Delaware
  - UM Sylvester Comprehensive Cancer Center at Coral Gables, Coral Gables, Florida
  - UM Sylvester Comprehensive Cancer Center at Deerfield Beach, Deerfield Beach, Florida
  - University of Florida Health Science Center - Gainesville, Gainesville, Florida
  - Mayo Clinic in Florida, Jacksonville, Florida
  - University of Miami Miller School of Medicine-Sylvester Cancer Center, Miami, Florida
  - Miami Cancer Institute, Miami, Florida
  - UM Sylvester Comprehensive Cancer Center at Kendall, Miami, Florida
  - Orlando Health Cancer Institute, Orlando, Florida
  - UM Sylvester Comprehensive Cancer Center at Plantation, Plantation, Florida
  - Tallahassee Memorial HealthCare, Tallahassee, Florida
  - Moffitt Cancer Center, Tampa, Florida
  - Cleveland Clinic-Weston, Weston, Florida
  - Grady Health System, Atlanta, Georgia
  - Emory University Hospital Midtown, Atlanta, Georgia
  - Emory University Hospital/Winship Cancer Institute, Atlanta, Georgia
  - Emory Saint Joseph's Hospital, Atlanta, Georgia
  - Augusta University Medical Center, Augusta, Georgia
  - Lewis Cancer and Research Pavilion at Saint Joseph's/Candler, Savannah, Georgia
  - Queen's Medical Center, Honolulu, Hawaii
  - The Cancer Center of Hawaii-Liliha, Honolulu, Hawaii
  - Saint Alphonsus Cancer Care Center-Nampa, Nampa, Idaho
  - Northwestern University, Chicago, Illinois
  - Rush University Medical Center, Chicago, Illinois
  - University of Illinois, Chicago, Illinois
  - Decatur Memorial Hospital, Decatur, Illinois
  - Crossroads Cancer Center, Effingham, Illinois
  - Western Illinois Cancer Treatment Center, Galesburg, Illinois
  - Edward Hines Jr VA Hospital, Hines, Illinois
  - Condell Memorial Hospital, Libertyville, Illinois
  - Loyola University Medical Center, Maywood, Illinois
  - Advocate Lutheran General Hospital, Park Ridge, Illinois
  - Methodist Medical Center of Illinois, Peoria, Illinois
  - OSF Saint Francis Medical Center, Peoria, Illinois
  - UW Health Carbone Cancer Center Rockford, Rockford, Illinois
  - Springfield Memorial Hospital, Springfield, Illinois
  - Southwest Illinois Health Services LLP, Swansea, Illinois
  - Carle Cancer Center, Urbana, Illinois
  - Parkview Hospital Randallia, Fort Wayne, Indiana
  - Parkview Regional Medical Center, Fort Wayne, Indiana
  - Goshen Center for Cancer Care, Goshen, Indiana
  - Community Cancer Center East, Indianapolis, Indiana
  - Community Cancer Center South, Indianapolis, Indiana
  - Franciscan Health Indianapolis, Indianapolis, Indiana
  - Community Cancer Center North, Indianapolis, Indiana
  - Franciscan Health Mooresville, Mooresville, Indiana
  - Mercy Cancer Center-West Lakes, Clive, Iowa
  - Iowa Methodist Medical Center, Des Moines, Iowa
  - Mercy Medical Center - Des Moines, Des Moines, Iowa
  - University of Kansas Cancer Center, Kansas City, Kansas
  - Lawrence Memorial Hospital, Lawrence, Kansas
  - University of Kansas Cancer Center-Overland Park, Overland Park, Kansas
  - Ascension Via Christi Hospitals Wichita, Wichita, Kansas
  - Saint Elizabeth Healthcare Edgewood, Edgewood, Kentucky
  - University of Kentucky/Markey Cancer Center, Lexington, Kentucky
  - Norton Hospital Pavilion and Medical Campus, Louisville, Kentucky
  - The James Graham Brown Cancer Center at University of Louisville, Louisville, Kentucky
  - Norton Brownsboro Hospital and Medical Campus, Louisville, Kentucky
  - LSU Health Baton Rouge-North Clinic, Baton Rouge, Louisiana
  - Our Lady of the Lake Physician Group, Baton Rouge, Louisiana
  - Louisiana Hematology Oncology Associates LLC, Baton Rouge, Louisiana
  - Mary Bird Perkins Cancer Center, Baton Rouge, Louisiana
  - University of Maryland/Greenebaum Cancer Center, Baltimore, Maryland
  - Central Maryland Radiation Oncology in Howard County, Columbia, Maryland
  - UM Baltimore Washington Medical Center/Tate Cancer Center, Glen Burnie, Maryland
  - TidalHealth Richard A Henson Cancer Institute, Ocean Pines, Maryland
  - TidalHealth Peninsula Regional, Salisbury, Maryland
  - Massachusetts General Hospital Cancer Center, Boston, Massachusetts
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Boston Medical Center, Boston, Massachusetts
  - Lahey Hospital and Medical Center, Burlington, Massachusetts
  - McLaren Cancer Institute-Bay City, Bay City, Michigan
  - McLaren Cancer Institute-Clarkston, Clarkston, Michigan
  - Henry Ford Macomb Hospital-Clinton Township, Clinton Township, Michigan
  - Wayne State University/Karmanos Cancer Institute, Detroit, Michigan
  - Henry Ford Hospital, Detroit, Michigan
  - Henry Ford Health Saint John Hospital, Detroit, Michigan
  - Weisberg Cancer Treatment Center, Farmington Hills, Michigan
  - McLaren Cancer Institute-Flint, Flint, Michigan
  - Singh and Arora Hematology Oncology PC, Flint, Michigan
  - Allegiance Health, Jackson, Michigan
  - West Michigan Cancer Center, Kalamazoo, Michigan
  - Karmanos Cancer Institute at McLaren Greater Lansing, Lansing, Michigan
  - Mid-Michigan Physicians-Lansing, Lansing, Michigan
  - University of Michigan Health - Sparrow Lansing, Lansing, Michigan
  - McLaren Cancer Institute-Lapeer Region, Lapeer, Michigan
  - Trinity Health Saint Mary Mercy Livonia Hospital, Livonia, Michigan
  - McLaren Cancer Institute-Macomb, Mount Clemens, Michigan
  - McLaren Cancer Institute-Northern Michigan, Petoskey, Michigan
  - Michigan Healthcare Professionals Pontiac, Pontiac, Michigan
  - McLaren-Port Huron, Port Huron, Michigan
  - Corewell Health William Beaumont University Hospital, Royal Oak, Michigan
  - MyMichigan Medical Center Saginaw, Saginaw, Michigan
  - Corewell Health Beaumont Troy Hospital, Troy, Michigan
  - Henry Ford Health Warren Hospital, Warren, Michigan
  - University of Michigan Health - West, Wyoming, Michigan
  - Sanford Joe Lueken Cancer Center, Bemidji, Minnesota
  - Saint Luke's Hospital of Duluth, Duluth, Minnesota
  - Hennepin County Medical Center, Minneapolis, Minnesota
  - Coborn Cancer Center at Saint Cloud Hospital, Saint Cloud, Minnesota
  - Regions Hospital, Saint Paul, Minnesota
  - Saint Francis Medical Center, Cape Girardeau, Missouri
  - Siteman Cancer Center at West County Hospital, Creve Coeur, Missouri
  - Kansas City Veterans Affairs Medical Center, Kansas City, Missouri
  - Delbert Day Cancer Institute at PCRMC, Rolla, Missouri
  - Mercy Hospital Springfield, Springfield, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Missouri Baptist Medical Center, St Louis, Missouri
  - Mercy Hospital Saint Louis, St Louis, Missouri
  - Bozeman Health Deaconess Hospital, Bozeman, Montana
  - Saint James Community Hospital and Cancer Treatment Center, Butte, Montana
  - Benefis Sletten Cancer Institute, Great Falls, Montana
  - Logan Health Medical Center, Kalispell, Montana
  - Nebraska Methodist Hospital, Omaha, Nebraska
  - Alegent Health Bergan Mercy Medical Center, Omaha, Nebraska
  - Renown Regional Medical Center, Reno, Nevada
  - Wentworth-Douglass Hospital, Dover, New Hampshire
  - Dartmouth Hitchcock Medical Center/Dartmouth Cancer Center, Lebanon, New Hampshire
  - Memorial Sloan Kettering Basking Ridge, Basking Ridge, New Jersey
  - Memorial Sloan Kettering Monmouth, Middletown, New Jersey
  - Memorial Sloan Kettering Bergen, Montvale, New Jersey
  - Virtua Samson Cancer Center, Moorestown, New Jersey
  - Virtua Memorial, Mount Holly, New Jersey
  - Community Medical Center, Toms River, New Jersey
  - Virtua Voorhees, Voorhees Township, New Jersey
  - Lovelace Medical Center-Saint Joseph Square, Albuquerque, New Mexico
  - University of New Mexico Cancer Center, Albuquerque, New Mexico
  - Lovelace Radiation Oncology, Albuquerque, New Mexico
  - Christus Saint Vincent Regional Cancer Center, Santa Fe, New Mexico
  - New York-Presbyterian/Brooklyn Methodist Hospital, Brooklyn, New York
  - Memorial Sloan Kettering Commack, Commack, New York
  - Memorial Sloan Kettering Westchester, East White Plains, New York
  - Mount Sinai West, New York, New York
  - Mount Sinai Hospital, New York, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - University of Rochester, Rochester, New York
  - Stony Brook University Medical Center, Stony Brook, New York
  - State University of New York Upstate Medical University, Syracuse, New York
  - Montefiore Medical Center-Einstein Campus, The Bronx, New York
  - Montefiore Medical Center - Moses Campus, The Bronx, New York
  - Memorial Sloan Kettering Nassau, Uniondale, New York
  - Dickstein Cancer Treatment Center, White Plains, New York
  - Carolinas Medical Center/Levine Cancer Institute, Charlotte, North Carolina
  - Atrium Health Pineville/LCI-Pineville, Charlotte, North Carolina
  - Atrium Health University City/LCI-University, Charlotte, North Carolina
  - Atrium Health Cabarrus/LCI-Concord, Concord, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - Atrium Health Union/LCI-Union, Monroe, North Carolina
  - CarolinaEast Medical Center, New Bern, North Carolina
  - Novant Cancer Institute Radiation Oncology - Supply, Supply, North Carolina
  - Novant Health Cancer Institute Radiation Oncology - Wilmington, Wilmington, North Carolina
  - Novant Health New Hanover Regional Medical Center, Wilmington, North Carolina
  - Sanford Bismarck Medical Center, Bismarck, North Dakota
  - Sanford Roger Maris Cancer Center, Fargo, North Dakota
  - Altru Cancer Center, Grand Forks, North Dakota
  - Cleveland Clinic Akron General, Akron, Ohio
  - UHHS-Chagrin Highlands Medical Center, Beachwood, Ohio
  - Geauga Hospital, Chardon, Ohio
  - Adena Regional Medical Center, Chillicothe, Ohio
  - University of Cincinnati Cancer Center-UC Medical Center, Cincinnati, Ohio
  - Case Western Reserve University, Cleveland, Ohio
  - Cleveland Clinic Cancer Center/Fairview Hospital, Cleveland, Ohio
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - The Mark H Zangmeister Center, Columbus, Ohio
  - Cleveland Clinic Cancer Center Mansfield, Mansfield, Ohio
  - Hillcrest Hospital Cancer Center, Mayfield Heights, Ohio
  - UH Seidman Cancer Center at Lake Health Mentor Campus, Mentor, Ohio
  - UH Seidman Cancer Center at Southwest General Hospital, Middleburg Heights, Ohio
  - University Hospitals Parma Medical Center, Parma, Ohio
  - University Hospitals Portage Medical Center, Ravenna, Ohio
  - North Coast Cancer Care, Sandusky, Ohio
  - UH Seidman Cancer Center at Firelands Regional Medical Center, Sandusky, Ohio
  - ProMedica Flower Hospital, Sylvania, Ohio
  - University of Cincinnati Cancer Center-West Chester, West Chester, Ohio
  - UH Seidman Cancer Center at Saint John Medical Center, Westlake, Ohio
  - UHHS-Westlake Medical Center, Westlake, Ohio
  - Cleveland Clinic Wooster Family Health and Surgery Center, Wooster, Ohio
  - Genesis Healthcare System Cancer Care Center, Zanesville, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Mercy Hospital Oklahoma City, Oklahoma City, Oklahoma
  - Good Samaritan Hospital, Corvallis, Oregon
  - Legacy Mount Hood Medical Center, Gresham, Oregon
  - Legacy Good Samaritan Hospital and Medical Center, Portland, Oregon
  - Providence Portland Medical Center, Portland, Oregon
  - Providence Saint Vincent Medical Center, Portland, Oregon
  - Bryn Mawr Hospital, Bryn Mawr, Pennsylvania
  - Geisinger Medical Center, Danville, Pennsylvania
  - Delaware County Memorial Hospital, Drexel Hill, Pennsylvania
  - Northeast Radiation Oncology Center, Dunmore, Pennsylvania
  - Saint Vincent Hospital, Erie, Pennsylvania
  - UPMC Pinnacle Cancer Center/Community Osteopathic Campus, Harrisburg, Pennsylvania
  - Penn State Milton S Hershey Medical Center, Hershey, Pennsylvania
  - Lancaster General Ann B Barshinger Cancer Institute, Lancaster, Pennsylvania
  - Lancaster General Hospital, Lancaster, Pennsylvania
  - Geisinger Medical Oncology-Lewisburg, Lewisburg, Pennsylvania
  - Lewistown Hospital, Lewistown, Pennsylvania
  - Paoli Memorial Hospital, Paoli, Pennsylvania
  - Thomas Jefferson University Hospital, Philadelphia, Pennsylvania
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - Jefferson Torresdale Hospital, Philadelphia, Pennsylvania
  - Geisinger Cancer Services-Pottsville, Pottsville, Pennsylvania
  - Guthrie Medical Group PC-Robert Packer Hospital, Sayre, Pennsylvania
  - Reading Hospital, West Reading, Pennsylvania
  - Geisinger Wyoming Valley/Henry Cancer Center, Wilkes-Barre, Pennsylvania
  - Asplundh Cancer Pavilion, Willow Grove, Pennsylvania
  - Lankenau Medical Center, Wynnewood, Pennsylvania
  - Prisma Health Cancer Institute - Spartanburg, Boiling Springs, South Carolina
  - Prisma Health Cancer Institute - Faris, Greenville, South Carolina
  - Saint Francis Cancer Center, Greenville, South Carolina
  - Prisma Health Cancer Institute - Eastside, Greenville, South Carolina
  - Self Regional Healthcare, Greenwood, South Carolina
  - Prisma Health Cancer Institute - Greer, Greer, South Carolina
  - Gibbs Cancer Center-Pelham, Greer, South Carolina
  - The Radiation Oncology Center-Hilton Head/Bluffton, Hilton Head Island, South Carolina
  - Prisma Health Cancer Institute - Seneca, Seneca, South Carolina
  - Spartanburg Medical Center, Spartanburg, South Carolina
  - Sanford USD Medical Center - Sioux Falls, Sioux Falls, South Dakota
  - Baptist Memorial Hospital and Cancer Center-Memphis, Memphis, Tennessee
  - UT Southwestern/Simmons Cancer Center-Dallas, Dallas, Texas
  - UT Southwestern/Simmons Cancer Center-Fort Worth, Fort Worth, Texas
  - University of Texas Medical Branch, Galveston, Texas
  - M D Anderson Cancer Center, Houston, Texas
  - Covenant Medical Center-Lakeside, Lubbock, Texas
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas
  - Huntsman Cancer Institute/University of Utah, Salt Lake City, Utah
  - George E Wahlen Department of Veterans Affairs Medical Center, Salt Lake City, Utah
  - Dartmouth Cancer Center - North, Saint Johnsbury, Vermont
  - VCU Massey Cancer Center at Stony Point, Richmond, Virginia
  - Virginia Commonwealth University/Massey Cancer Center, Richmond, Virginia
  - Legacy Salmon Creek Hospital, Vancouver, Washington
  - West Virginia University Healthcare, Morgantown, West Virginia
  - Langlade Hospital and Cancer Center, Antigo, Wisconsin
  - Ascension Saint Elizabeth Hospital, Appleton, Wisconsin
  - Aurora Cancer Care-Southern Lakes VLCC, Burlington, Wisconsin
  - Marshfield Medical Center-EC Cancer Center, Eau Claire, Wisconsin
  - Aurora Health Center-Fond du Lac, Fond du Lac, Wisconsin
  - Aurora Health Care Germantown Health Center, Germantown, Wisconsin
  - Aurora Cancer Care-Grafton, Grafton, Wisconsin
  - Saint Vincent Hospital Cancer Center Green Bay, Green Bay, Wisconsin
  - Saint Vincent Hospital Cancer Center at Saint Mary's, Green Bay, Wisconsin
  - Aurora BayCare Medical Center, Green Bay, Wisconsin
  - Aurora Cancer Care-Kenosha South, Kenosha, Wisconsin
  - Gundersen Lutheran Medical Center, La Crosse, Wisconsin
  - Aurora Bay Area Medical Group-Marinette, Marinette, Wisconsin
  - Marshfield Medical Center-Marshfield, Marshfield, Wisconsin
  - Froedtert Menomonee Falls Hospital, Menomonee Falls, Wisconsin
  - Aurora Cancer Care-Milwaukee, Milwaukee, Wisconsin
  - Aurora Saint Luke's Medical Center, Milwaukee, Wisconsin
  - Medical College of Wisconsin, Milwaukee, Wisconsin
  - Aurora Sinai Medical Center, Milwaukee, Wisconsin
  - Marshfield Medical Center - Minocqua, Minocqua, Wisconsin
  - Ascension Mercy Hospital, Oshkosh, Wisconsin
  - Vince Lombardi Cancer Clinic - Oshkosh, Oshkosh, Wisconsin
  - Aurora Cancer Care-Racine, Racine, Wisconsin
  - Vince Lombardi Cancer Clinic-Sheboygan, Sheboygan, Wisconsin
  - Marshfield Medical Center-River Region at Stevens Point, Stevens Point, Wisconsin
  - Aurora Medical Center in Summit, Summit, Wisconsin
  - Vince Lombardi Cancer Clinic-Two Rivers, Two Rivers, Wisconsin
  - Aspirus Regional Cancer Center, Wausau, Wisconsin
  - Aurora Cancer Care-Milwaukee West, Wauwatosa, Wisconsin
  - Aurora West Allis Medical Center, West Allis, Wisconsin
  - Froedtert West Bend Hospital/Kraemer Cancer Center, West Bend, Wisconsin
  - Marshfield Medical Center - Weston, Weston, Wisconsin
  - Aspirus Cancer Care - Wisconsin Rapids, Wisconsin Rapids, Wisconsin
- Canada (3):
  - Cross Cancer Institute, Edmonton, Alberta
  - London Regional Cancer Program, London, Ontario
  - Ottawa Hospital and Cancer Center-General Campus, Ottawa, Ontario
- Chaim Sheba Medical Center, Tel Litwinsky, Israel
- King Faisal Specialist Hospital and Research Centre, Riyadh, Saudi Arabia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Mattes MD, Eubank TD, Almubarak M, Wen S, Marano GD, Jacobson GM, Ma PC. A Prospective Trial Evaluating the Safety and Systemic Response From the Concurrent Use of Radiation Therapy with Checkpoint Inhibitor Immunotherapy in Metastatic Non-Small Cell Lung Cancer. Clin Lung Cancer. 2021 Jul;22(4):268-273. doi: 10.1016/j.cllc.2021.01.012. Epub 2021 Jan 25. PMID 33608212

RESULTS

PARTICIPANT FLOW:
Groups:
- Arm 2 (LCT + systemic maintenance chemotherapy): Patients undergo local consolidative therapy (LCT) over 2-5 weeks, consisting of stereotactic body radiation therapy (SBRT)/hypofractionated radiation to the primary tumor and metastatic sites or surgery of metastatic sites. Hypofractionated radiation using intensity modulated radiation therapy (IMRT) or 3-dimensional conformal radiation therapy (3D-CRT) can be given in place of SBRT. Within 2 weeks after completion of LCT (3 weeks if surgery occurred), patients receive chemotherapy as in Arm 1.
Period: Overall Study
Arm/Group | Arm 1 (systemic maintenance chemotherapy) | Arm 2 (LCT + systemic maintenance chemotherapy)
Started | 82 | 136
Modified intent-to-treat (MITT) population (Randomized and eligible.) | 81 | 134
Completed (Patients contributing data to any results are considered to have completed the study.) | 81 | 134
Not Completed | 1 | 2

BASELINE CHARACTERISTICS:
Population: Modified intent-to-treat population (randomized and eligible).
Groups:
- Arm 2 (LCT + Systemic Maintenance Chemotherapy): Patients undergo local consolidative therapy (LCT) over 2-5 weeks, consisting of SBRT/hypofractionated radiation to the primary tumor and metastatic sites or surgery of metastatic sites. Hypofractionated radiation using IMRT or 3DCRT can be given in place of SBRT. Within 2 weeks after completion of LCT (3 weeks if surgery occurred), patients receive chemotherapy as in Arm 1.
- Total: Total of all reporting groups
Arm/Group | Arm 1 (Systemic Maintenance Chemotherapy) | Arm 2 (LCT + Systemic Maintenance Chemotherapy) | Total
Number analyzed (Participants) | 81 | 134 | 215
Age, Customized [Count of Participants; unit: Participants]
  ≤ 49 years | 4 | 4 | 8
  50 - 59 years | 15 | 29 | 44
  60 - 69 years | 31 | 56 | 87
  ≥ 70 years | 31 | 45 | 76
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 41 | 66 | 107
  Male | 40 | 68 | 108
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 7 | 9
  Not Hispanic or Latino | 78 | 118 | 196
  Unknown or Not Reported | 1 | 9 | 10
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 1 | 2
  Asian | 2 | 2 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 16 | 19 | 35
  White | 59 | 106 | 165
  More than one race | 1 | 0 | 1
  Unknown or Not Reported | 2 | 6 | 8
Zubrod performance status [Count of Participants; unit: Participants] — 0 = Asymptomatic; 1 = Symptomatic but completely ambulatory; 2 = Symptomatic, <50% in bed during the day; 3 = Symptomatic, >50% in bed, but not bedbound; 4 = Bedbound; 5 = Death.
  Participants
    0 | 35 | 47 | 82
    1 | 44 | 79 | 123
    2 | 2 | 8 | 10
Histology [Count of Participants; unit: Participants] — A description of a tumor based on how the cancer cells and tissue look under a microscope.
  Participants
    Non-Squamous cell carcinoma | 64 | 104 | 168
    Squamous cell carcinoma | 17 | 30 | 47
Systemic Therapy Type [Count of Participants; unit: Participants]
  Cytotoxic Chemotherapy | 14 | 16 | 30
  Immunotherapy | 67 | 118 | 185
Number of lesions targeted during treatment [Count of Participants; unit: Participants]
  1 | 50 | 78 | 128
  2 | 19 | 36 | 55
  3 | 12 | 18 | 30
  4 | 0 | 1 | 1
  5 | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: [Phase II] Progression-free Survival
Description: Progression-free survival (PFS) is estimated by the Kaplan-Meier method. Progression-free survival time is measured from randomization to the first date of local or regional disease, distant metastases, second primary tumor, death due to any cause, or last known follow-up (censored). Analysis was to occur after progression or death was reported for 138 participants.
Time Frame: From randomization to first date of local or regional disease, distant metastases, second primary tumor, death, or last follow-up, whichever comes first. Maximum follow-up time at time of analysis was 5.4 years.
Population: Modified intent-to-treat population (randomized eligible participants).
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm 1 (systemic maintenance chemotherapy) | Arm 2 (LCT + systemic maintenance chemotherapy)
Number analyzed (Participants) | 81 | 134
months | 11.1 [6.9 to 21.4] | 13.7 [8.6 to 20.1]
Statistical Analysis 1: Comparison: Arm 1 (systemic maintenance chemotherapy) vs Arm 2 (LCT + systemic maintenance chemotherapy); Based on expected 6- and 12-month PFS rates of approximately 60% and 39% for the standard arm, assuming approximately exponential distributions, at least 138 PFS events are needed to detect a hazard ratio of 0.6 (a hazard reduction of 40%) with 95% power and a one-sided significance level of 0.15. The Cox proportional hazards model is stratified by histology and systemic therapy type. The hazard ratio estimate must be ≤ 0.83 for the study to proceed to the phase III component; Test type: Superiority; p = 0.66, Log Rank; Two-sided test; Hazard Ratio (HR) = 0.98, 95% CI 2-sided [0.68 to 1.40] — Reference level = systemic therapy. Cox proportional hazards model stratified by histology (non-squamous vs squamous) and systemic therapy (immunotherapy-based regimens vs chemotherapy- only regimens)

2. Primary Outcome: [Phase III] Overall Survival
Description: Overall survival is estimated by the Kaplan-Meier method. Survival time is measured from randomization to date of death from any cause or last known follow-up (censored). Analysis was to occur after **** deaths were reported.
Time Frame: From randomization to death or last follow-up.
Population: The phase III component did not open, therefore there are no participants for this outcome measure.
Arm/Group | Arm 1 (systemic maintenance chemotherapy) | Arm 2 (LCT + systemic maintenance chemotherapy)
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: In-Field Local Failure
Description: In-field local failure is defined as local or marginal failure. In-field local failure rates are estimated by the cumulative incidence method, in which death without failure is treated as competing risk and participants alive without failure are censored at last known follow-up. Analysis was to occur after progression or death was reported for 138 participants.
Time Frame: From randomization to first in-field failure, death or last follow-up, whichever occurs first. Maximum follow-up at time of analysis was 5.4 years. The one- and two-year estimates are reported.
Population: Modified intent-to-treat population (randomized eligible participants).
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Arm 1 (systemic maintenance chemotherapy) | Arm 2 (LCT + systemic maintenance chemotherapy)
Number analyzed (Participants) | 81 | 134
percentage of participants
  1 year | 15.3 [8.1 to 24.6] | 8.6 [4.6 to 14.3]
  2 years | 19.8 [11.4 to 29.9] | 13.4 [8.1 to 20.0]

4. Secondary Outcome: Development of New Lesions
Description: New lesion rates are estimated by the cumulative incidence method, in which death without new lesions is treated as competing risk and participants alive without new lesions are censored at last known follow-up. Analysis was to occur after progression or death was reported for 138 participants.
Time Frame: From randomization to the first occurrence of any new lesions, death, or last follow-up, whichever occurs first. Maximum follow-up time at the time of analysis was 5.4 years. One- and two-year estimates are reported.
Population: Modified intent-to-treat population (randomized eligible participants).
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Arm 1 (systemic maintenance chemotherapy) | Arm 2 (LCT + systemic maintenance chemotherapy)
Number analyzed (Participants) | 81 | 134
percentage of participants
  1 year | 32.5 [21.8 to 43.5] | 28.1 [20.6 to 36.1]
  2 years | 41.5 [29.7 to 52.9] | 30.5 [22.7 to 38.6]

5. Secondary Outcome: Number of Participants by Highest Grade Adverse Event Reported
Description: National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version 5.0 grades adverse event severity as follows: 1 = mild, 2 = moderate, 3 = severe, 4 = life-threatening, 5 = death related to adverse event. Summary data is provided in this outcome measure; see Adverse Events Module for specific adverse event data.
Time Frame: From randomization to last follow-up. Maximum follow-up at time of analysis was 5.4 years.
Population: Modified intent-to-treat population (randomized and eligible) who received any protocol treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 1 (systemic maintenance chemotherapy) | Arm 2 (LCT + systemic maintenance chemotherapy)
Number analyzed (Participants) | 73 | 130
Participants
  Grade 1 | 7 | 6
  Grade 2 | 15 | 37
  Grade 3 | 35 | 56
  Grade 4 | 11 | 20
  Grade 5 | 4 | 10
  None | 1 | 1

6. Secondary Outcome: Duration of Maintenance Chemotherapy
Description: Duration of Maintenance Chemotherapy
Time Frame: From randomization to last chemotherapy, which continues until progression or significant toxicity. Maximum follow-up at time of analysis was 5.4 years.
Population: Modified intent-to-treat population (randomized eligible participants).
Measure: Median (Inter-Quartile Range); unit: months
Arm/Group | Arm 1 (systemic maintenance chemotherapy) | Arm 2 (LCT + systemic maintenance chemotherapy)
Number analyzed (Participants) | 81 | 134
months | 5.46 [2.07 to 17.95] | 6.20 [2.81 to 16.86]

ADVERSE EVENTS:
Time Frame: From baseline to date of last known follow-up. Maximum follow-up time was 5.4 years.
Description: All-cause mortality was assessed in the modified intent-to-treat population (MITT) (randomized and eligible). Adverse events were assessed in the MITT population that started protocol treatment.
Arm/Group | Arm 1 (systemic maintenance chemotherapy) | Arm 2 (LCT + systemic maintenance chemotherapy)
All-Cause Mortality (participants affected / at risk) | 37/81 | 70/134
Serious Adverse Events (participants affected / at risk) | 14/73 | 40/130
Other Adverse Events (participants affected / at risk) | 71/73 | 129/130
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm 1 (systemic maintenance chemotherapy) (N=73) | Arm 2 (LCT + systemic maintenance chemotherapy) (N=130)
Anemia (Blood and lymphatic system disorders) | 0 | 3
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 1
Cardiac arrest (Cardiac disorders) | 1 | 0
Cardiac disorders - Other (Cardiac disorders) | 0 | 1
Chest pain - cardiac (Cardiac disorders) | 0 | 1
Myocardial infarction (Cardiac disorders) | 0 | 3
Pericardial effusion (Cardiac disorders) | 1 | 0
Pericarditis (Cardiac disorders) | 0 | 1
Sinus tachycardia (Cardiac disorders) | 0 | 1
Hypophysitis (Endocrine disorders) | 0 | 1
Colitis (Gastrointestinal disorders) | 0 | 1
Colonic perforation (Gastrointestinal disorders) | 0 | 1
Diarrhea (Gastrointestinal disorders) | 0 | 1
Esophageal pain (Gastrointestinal disorders) | 0 | 1
Esophagitis (Gastrointestinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 0 | 1
Death NOS (General disorders and administration site conditions) | 0 | 2
Disease progression (General disorders and administration site conditions) | 0 | 1
Fatigue (General disorders and administration site conditions) | 0 | 1
Malaise (General disorders and administration site conditions) | 0 | 1
Sudden death NOS (General disorders and administration site conditions) | 1 | 0
Cholecystitis (Hepatobiliary disorders) | 0 | 1
Cytomegalovirus infection reactivation (Infections and infestations) | 0 | 1
Encephalitis infection (Infections and infestations) | 0 | 1
Herpes simplex reactivation (Infections and infestations) | 0 | 1
Lung infection (Infections and infestations) | 1 | 6
Sepsis (Infections and infestations) | 0 | 3
Fall (Injury, poisoning and procedural complications) | 0 | 1
Injury, poisoning and procedural complications - Other (Injury, poisoning and procedural complications) | 0 | 1
Postoperative hemorrhage (Injury, poisoning and procedural complications) | 0 | 1
Alkaline phosphatase increased (Investigations) | 1 | 0
Aspartate aminotransferase increased (Investigations) | 1 | 0
Ejection fraction decreased (Investigations) | 0 | 1
Neutrophil count decreased (Investigations) | 0 | 1
White blood cell decreased (Investigations) | 0 | 1
Acidosis (Metabolism and nutrition disorders) | 0 | 1
Anorexia (Metabolism and nutrition disorders) | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 2
Hyperglycemia (Metabolism and nutrition disorders) | 0 | 1
Hyponatremia (Metabolism and nutrition disorders) | 0 | 1
Metabolism and nutrition disorders - Other (Metabolism and nutrition disorders) | 0 | 1
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 0 | 1
Cognitive disturbance (Nervous system disorders) | 1 | 0
Ischemia cerebrovascular (Nervous system disorders) | 0 | 1
Peripheral sensory neuropathy (Nervous system disorders) | 0 | 1
Seizure (Nervous system disorders) | 2 | 0
Stroke (Nervous system disorders) | 0 | 1
Confusion (Psychiatric disorders) | 0 | 1
Acute kidney injury (Renal and urinary disorders) | 1 | 1
Urinary incontinence (Renal and urinary disorders) | 0 | 1
Urinary tract obstruction (Renal and urinary disorders) | 0 | 1
Bronchial obstruction (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 | 5
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 3
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 2 | 7
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 5
Respiratory, thoracic and mediastinal disorders - Other (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 | 1
Arterial thromboembolism (Vascular disorders) | 0 | 1
Hypotension (Vascular disorders) | 0 | 1
Thromboembolic event (Vascular disorders) | 1 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Arm 1 (systemic maintenance chemotherapy) (N=73) | Arm 2 (LCT + systemic maintenance chemotherapy) (N=130)
Anemia (Blood and lymphatic system disorders) | 34 | 67
Blood and lymphatic system disorders - Other (Blood and lymphatic system disorders) | 5 | 4
Atrial fibrillation (Cardiac disorders) | 0 | 8
Cardiac disorders - Other (Cardiac disorders) | 4 | 5
Sinus tachycardia (Cardiac disorders) | 2 | 10
Hearing impaired (Ear and labyrinth disorders) | 6 | 10
Hyperthyroidism (Endocrine disorders) | 6 | 2
Hypothyroidism (Endocrine disorders) | 15 | 14
Blurred vision (Eye disorders) | 7 | 12
Dry eye (Eye disorders) | 8 | 5
Eye disorders - Other (Eye disorders) | 10 | 6
Eye pain (Eye disorders) | 5 | 2
Watering eyes (Eye disorders) | 6 | 3
Abdominal pain (Gastrointestinal disorders) | 13 | 24
Constipation (Gastrointestinal disorders) | 22 | 34
Diarrhea (Gastrointestinal disorders) | 22 | 33
Dry mouth (Gastrointestinal disorders) | 7 | 6
Dyspepsia (Gastrointestinal disorders) | 8 | 9
Dysphagia (Gastrointestinal disorders) | 4 | 22
Esophagitis (Gastrointestinal disorders) | 1 | 22
Gastroesophageal reflux disease (Gastrointestinal disorders) | 5 | 12
Gastrointestinal disorders - Other (Gastrointestinal disorders) | 7 | 10
Mucositis oral (Gastrointestinal disorders) | 5 | 13
Nausea (Gastrointestinal disorders) | 31 | 46
Vomiting (Gastrointestinal disorders) | 15 | 26
Chills (General disorders and administration site conditions) | 4 | 17
Edema face (General disorders and administration site conditions) | 5 | 6
Edema limbs (General disorders and administration site conditions) | 19 | 25
Fatigue (General disorders and administration site conditions) | 42 | 91
Fever (General disorders and administration site conditions) | 9 | 20
Gait disturbance (General disorders and administration site conditions) | 8 | 7
General disorders and administration site conditions - Other (General disorders and administration site conditions) | 8 | 11
Localized edema (General disorders and administration site conditions) | 5 | 12
Non-cardiac chest pain (General disorders and administration site conditions) | 8 | 20
Pain (General disorders and administration site conditions) | 8 | 17
Infections and infestations - Other (Infections and infestations) | 8 | 17
Lung infection (Infections and infestations) | 5 | 23
Sepsis (Infections and infestations) | 3 | 7
Skin infection (Infections and infestations) | 4 | 2
Upper respiratory infection (Infections and infestations) | 4 | 8
Urinary tract infection (Infections and infestations) | 6 | 12
Bruising (Injury, poisoning and procedural complications) | 4 | 9
Fall (Injury, poisoning and procedural complications) | 12 | 11
Injury, poisoning and procedural complications - Other (Injury, poisoning and procedural complications) | 7 | 4
Alanine aminotransferase increased (Investigations) | 15 | 24
Alkaline phosphatase increased (Investigations) | 9 | 19
Aspartate aminotransferase increased (Investigations) | 16 | 20
Blood bilirubin increased (Investigations) | 4 | 4
Cholesterol high (Investigations) | 4 | 5
Creatinine increased (Investigations) | 20 | 34
Investigations - Other (Investigations) | 6 | 14
Lymphocyte count decreased (Investigations) | 16 | 57
Neutrophil count decreased (Investigations) | 7 | 16
Platelet count decreased (Investigations) | 11 | 26
Thyroid stimulating hormone increased (Investigations) | 8 | 6
Weight gain (Investigations) | 5 | 7
Weight loss (Investigations) | 13 | 25
White blood cell decreased (Investigations) | 9 | 31
Anorexia (Metabolism and nutrition disorders) | 19 | 38
Dehydration (Metabolism and nutrition disorders) | 2 | 12
Hypercalcemia (Metabolism and nutrition disorders) | 8 | 18
Hyperglycemia (Metabolism and nutrition disorders) | 26 | 35
Hyperkalemia (Metabolism and nutrition disorders) | 9 | 16
Hypoalbuminemia (Metabolism and nutrition disorders) | 18 | 22
Hypocalcemia (Metabolism and nutrition disorders) | 9 | 11
Hypokalemia (Metabolism and nutrition disorders) | 18 | 33
Hypomagnesemia (Metabolism and nutrition disorders) | 3 | 9
Hyponatremia (Metabolism and nutrition disorders) | 22 | 31
Arthralgia (Musculoskeletal and connective tissue disorders) | 9 | 17
Arthritis (Musculoskeletal and connective tissue disorders) | 5 | 14
Back pain (Musculoskeletal and connective tissue disorders) | 16 | 32
Bone pain (Musculoskeletal and connective tissue disorders) | 5 | 6
Chest wall pain (Musculoskeletal and connective tissue disorders) | 2 | 9
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 10 | 10
Muscle cramp (Musculoskeletal and connective tissue disorders) | 4 | 4
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 1 | 8
Musculoskeletal and connective tissue disorder - Other (Musculoskeletal and connective tissue disorders) | 8 | 14
Myalgia (Musculoskeletal and connective tissue disorders) | 15 | 19
Neck pain (Musculoskeletal and connective tissue disorders) | 6 | 17
Pain in extremity (Musculoskeletal and connective tissue disorders) | 15 | 14
Concentration impairment (Nervous system disorders) | 4 | 2
Dizziness (Nervous system disorders) | 16 | 32
Dysesthesia (Nervous system disorders) | 5 | 3
Dysgeusia (Nervous system disorders) | 7 | 12
Headache (Nervous system disorders) | 20 | 27
Memory impairment (Nervous system disorders) | 7 | 12
Paresthesia (Nervous system disorders) | 10 | 11
Peripheral motor neuropathy (Nervous system disorders) | 6 | 3
Peripheral sensory neuropathy (Nervous system disorders) | 13 | 24
Tremor (Nervous system disorders) | 1 | 9
Anxiety (Psychiatric disorders) | 11 | 13
Confusion (Psychiatric disorders) | 10 | 4
Depression (Psychiatric disorders) | 11 | 14
Insomnia (Psychiatric disorders) | 10 | 25
Chronic kidney disease (Renal and urinary disorders) | 1 | 8
Dysuria (Renal and urinary disorders) | 4 | 4
Proteinuria (Renal and urinary disorders) | 4 | 6
Renal and urinary disorders - Other (Renal and urinary disorders) | 4 | 5
Urinary frequency (Renal and urinary disorders) | 4 | 8
Urinary incontinence (Renal and urinary disorders) | 5 | 4
Urinary urgency (Renal and urinary disorders) | 1 | 8
Pelvic pain (Reproductive system and breast disorders) | 4 | 2
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 10 | 9
Cough (Respiratory, thoracic and mediastinal disorders) | 20 | 49
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 27 | 63
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 4 | 8
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 2 | 8
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 6 | 23
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 11 | 19
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 3 | 14
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 11 | 24
Productive cough (Respiratory, thoracic and mediastinal disorders) | 10 | 35
Respiratory, thoracic and mediastinal disorders - Other (Respiratory, thoracic and mediastinal disorders) | 5 | 10
Sleep apnea (Respiratory, thoracic and mediastinal disorders) | 4 | 1
Sore throat (Respiratory, thoracic and mediastinal disorders) | 3 | 10
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 | 15
Alopecia (Skin and subcutaneous tissue disorders) | 6 | 7
Dry skin (Skin and subcutaneous tissue disorders) | 7 | 6
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 6 | 10
Pruritus (Skin and subcutaneous tissue disorders) | 10 | 21
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 9 | 13
Skin and subcutaneous tissue disorders - Other (Skin and subcutaneous tissue disorders) | 12 | 19
Hot flashes (Vascular disorders) | 5 | 5
Hypertension (Vascular disorders) | 24 | 31
Hypotension (Vascular disorders) | 4 | 17

LIMITATIONS AND CAVEATS:
Per the planned protocol analysis after the phase II component, the study did not proceed to the phase III component.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
PI's are required to abide by the sponsor's publication guidelines which require review by coauthors and subsequent review and approval by the sponsor.

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-10-18): https://cdn.clinicaltrials.gov/large-docs/71/NCT03137771/Prot_SAP_000.pdf
  • Informed Consent Form (2023-10-18): https://cdn.clinicaltrials.gov/large-docs/71/NCT03137771/ICF_001.pdf